CLINICAL TRIAL: NCT04028999
Title: Implementation of Supportive Sling Device in Adults Post-stroke for Prevention of Shoulder Complications
Acronym: EO31
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0460
Record Dates: First submitted 2019-07-11; First posted 2019-07-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cerebrovascular Accident
Keywords: Cerebrovascular Accident; sling; Upper limb impairment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the EO31 shoulder sling (Experimental): To develop and evaluate the effects of the EO31 shoulder sling for the prevention of pain, subluxation, spasticity, as well as effect on increasing functional use of the UL in activities of daily living.
  Interventions: Device: Evaluate the effects of the EO31 shoulder sling in adults post-stoke

INTERVENTIONS:
Device: Evaluate the effects of the EO31 shoulder sling in adults post-stoke — Investigator want to evaluate the efficient of the EO31 shoulder sling in adults post-stroke. The EO31 shoulder sling is made-to-measure shoulder pads for upper limb after cerebrovascular accident

SUMMARY:
Upper limb (UL) impairment is a common deficit following stroke with only an estimated 20 per cent of patients recovering function.

DETAILED DESCRIPTION:
Upper limb (UL) impairment is a common deficit following stroke with only an estimated 20 per cent of patients recovering function. Pain associated with UL impairment due to multifactorial causes is a frequent symptom in patients with stroke. Occupational therapy techniques focus on the implementation of positioning techniques and the use of supportive devices (SD) such as slings aimed to prevent pain; therefore increase daily function, participation and hence quality of life. At present, positioning principles of the hemiplegic shoulder exist in clinical practice. These are aimed at prevention of pain associated with UL Impairment; however there is no clear consensus among professionals of particular SD that should be implemented for adults with stroke

ELIGIBILITY:
Inclusion Criteria:

* Having suffered in the last 6 months maximum a first stroke responsible for hemiplegia.
* Finding a clinical 5mm appendix, or with shoulder pain requiring prescription a scarf.
* Boston Diagnostic Aphasia Examination (BDAE) > 3.
* Consent of the patient
* Patient affiliated or benefiting from a social security scheme

Exclusion Criteria:

* Stroke recurrence, or stroke more than 6 months-old
* Patient already wearing a coaptation scarf
* Presence of lymphoedema, venous thrombosis of the upper limb
* Neoprene allergy
* Severe cognitive impairment: Mini-Mental State (MMS) <15
* Patient being part of another care protocol
* Adult under the protection of justice, tutors or curators
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of the EO31 shoulder with Goal Attainment Scale (GAS) scale | 5 weeks
  GAS (Goal Attainment Scale) scores will be described with regards to the 3 client-centred objectives. The score for each objective is comprised between -2 (when objective is not achieve) to 2 (achieve objective).

SECONDARY OUTCOMES:
Evaluate shoulder pain with Visual Analog Scale for Pain (EVA scale) | 24 hours
  The shoulder pain will be evaluate with th sling with EVA Scale. Eva scale is between 0 (no pain) to 10 (big pain)
Evaluate shoulder pain with EVA scale | 5 weeks
  The shoulder pain will be evaluate with th sling with EVA Scale. Eva scale is between 0 (no pain) to 10 (big pain).
Evaluate shoulder pain with EVA scale | baseline
  The shoulder pain will be evaluate with th sling with EVA Scale. Eva scale is between 0 (no pain) to 10 (big pain).
Spasticity with TARDIEU scale | baseline
  Evaluate the spasticity of upper limb with TARDIEU scale: the rotation angle of the shoulder, elbow and wrist are measured
Spasticity with TARDIEU scale | 7 days
  Evaluate the spasticity of upper limb with TARDIEU scale: the rotation angle of the shoulder, elbow and wrist are measured
Spasticity with TARDIEU scale | 14 days
  Evaluate the spasticity of upper limb with TARDIEU scale: the rotation angle of the shoulder, elbow and wrist are measured
Spasticity with TARDIEU scale | 5 weeks
  Evaluate the spasticity of upper limb with TARDIEU scale: the rotation angle of the shoulder, elbow and wrist are measured
Number of daily use of the upper limb sling | 5 weeks
  Evaluate if patient use the sling : number of use by day
Clinical measure of appendage | baseline
  Evaluate of appendage with clinical measure during all the treatment. This measure is in millimeter
Clinical measure of appendage | 7 days
  Evaluate of appendage with clinical measure during all the treatment. This measure is in millimeter
Clinical measure of appendage | 14 days
  Evaluate of appendage with clinical measure during all the treatment. This measure is in millimeter
Clinical measure of appendage | 5 weeks
  Evaluate of appendage with clinical measure during all the treatment. This measure is in millimeter.
motor function of upper limb with Chedoke Arm and Hand Activity Inventory (CAHAI) scale | baseline
  the motor function of the upper limb will be evaluate with CAHAI scale between 13 (motor function low) to 94 (motor function strong)
motor function of upper limb with CAHAI scale | 7 days
  the motor function of the upper limb will be evaluate with CAHAI scale between 13 (motor function low) to 94 (motor function strong)
motor function of upper limb with CAHAI scale | 5 weeks
  the motor function of the upper limb will be evaluate with CAHAI scale between 13 (motor function low) to 94 (motor function strong)
questionnaire for quality of patient's life | baseline
  the quality of patient's life will be evaluate with ESAT scale between 0 (quality of life low) and 60 (good quality of life)
questionnaire for quality of patient's life | 5 weeks
  the quality of patient's life will be evaluate with ESAT scale between 0 (quality of life low) and 60 (good quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Castel-Lacanal, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montane E, Pradie M, Bigarre I, Lebely C, Lelievre A, Cormier C, Butterworth J, Lepage B, Marque P, de Boissezon X, Castel-Lacanal E. A custom-made sling to achieve personal goals in shoulder pain or subluxation in the subacute stroke phase: a pilot study. Ann Phys Rehabil Med. 2025 Oct;68(7):102014. doi: 10.1016/j.rehab.2025.102014. Epub 2025 Aug 21. PMID 40845630